CLINICAL TRIAL: NCT05720299
Title: A Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate the Effects of Akkermansia Muciniphila and Berberine on Prediabetes Among Obese Subjects.
Brief Title: A Clinical Study to Evaluate the Effects of Akkermansia Muciniphila and Berberine on Prediabetes Among Obese Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yu Chen (Other)
Responsible Party: Sponsor-Investigator, Yu Chen, Chief of Department of Gastroenterology, The Seventh Affiliated Hospital, Southern Medical University
Organization: The Seventh Affiliated Hospital, Southern Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZY19-202201
Record Dates: First submitted 2022-11-07; First posted 2023-02-09 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Prediabetes
Keywords: Akkermania muciniphila; obesity; metabolism; fecal flora; Prediabetes
MeSH Terms: conditions — Prediabetic State; Obesity | interventions — Berberine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Akkermansia muciniphila group(AKK) (Experimental): They will be treated with one tablet of AKK, twice a day, for 12 weeks.
  Interventions: Drug: Akkermansia muciniphila
- Berberine group (Experimental): They will be treated with one tablet of Berberine, twice a day, for 12 weeks.
  Interventions: Drug: Berberine
- Placebo group (Placebo Comparator): They will be treated with one tablet of placebo, twice a day, for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Akkermansia muciniphila — one tablet of AKK
  Arms: Akkermansia muciniphila group(AKK)
Drug: Berberine — one tablet of Berberine
  Arms: Berberine group
Drug: Placebo — one tablet of placebo
  Arms: Placebo group

SUMMARY:
The Akkermania muciniphila may play an important role in the occurrence and development of Prediabetes. The purpose of this study was to evaluate the safety and efficacy of AKK in the treatment of Prediabetes among obese patients. In this study, a single center, randomized, double-blind, placebo-controlled design is adopted. 90 obese subjects with Prediabetes are included in this study, and are allocated to AKK group, BBR group, and placebo group at a ratio of 1:1:1. The study treatment lasts for 12 weeks. The changes of body fat, glucose metabolism, lipid metabolism indicators compared with the baseline at the end of the treatment will be analyzed. In addition, glucagon like peptide-1 (GLP-1) and inflammatory markers (hsCRP、TNF-α、IL-6、IL-8、IL-1β) in blood will be analyzed before and after treatment. The changes in fecal flora structure and the AKK bacteria also will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65
2. Overweight/obesity (24.0≤BMI≤40.0 kg/m^2)
3. Fasting blood glucose ≥6.1 and <7.0 mmol/L, or 2-hour postprandial blood glucose ≥7.8 and <11.1 mmol/L, or glycosylated hemoglobin ≥5.7% and <6.5%
4. Fertile subjects (including male and female subjects) agreed to take effective contraceptive measures that the investigator accepted during and within 3 months after the trial (e.g. intrauterine device or a condom); the fertile female subjects with serum human chorionic gonadotropin test negative results within 7 days before the investigational product administration; Infertile female must be surgically infertile or at least 1 year after menopause.
5. Subjects should understand the nature, significance, potential benefits, inconvenience and risks of the study before the trial begins, fully understand and voluntarily sign the informed consent.

Exclusion Criteria:

1. Subjects who diagnosed with diabetes mellitus, medical obesity (excluding those who have been off medication for more than 1 year), or other secondary diabetes mellitus (e.g., Cushing's syndrome, thyroid dysfunction, or acromegaly);
2. Subjects who has undergone bariatric surgery;
3. Subjects who has acute or chronic progressive or unstable disease, liver and kidney insufficiency, serious cardiovascular and cerebrovascular diseases;

3.Subjects with acute diabetic complications such as diabetic ketoacidosis or diabetic hypertonic coma within within latest 3 months; 4.Patients with hemolytic anemia or glucose-6-phosphate dehydrogenase deficiency; 5.History of intestinal or intestinal surgery within 1 year, or non-gastrointestinal surgery within 6 months; 6.Excessive alcohol consumption in the last 10 years (more than 30 g/ day for male and 20g/ day for female) 7.Pregnant or lactating subjects 8.Subjects that the investigator considers need to excluded due to other causes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
HbA1c after 12weeks | Baseline , Day84
  Change from baseline in HbA1c

SECONDARY OUTCOMES:
Weight after 12weeks | Baseline , Day84
  Change from baseline in weight
Fasting and OGTT 2h blood glucose levels after 12weeks | Baseline , Day84
  Change from baseline in Fasting and OGTT 2h blood glucose levels
HOMA-IR after 12weeks | Baseline , Day84
  Change from baseline in HOMA-IR
Fasting and OGTT 2h insulin and C-peptide levels after 12weeks | Baseline , Day84
  Change from baseline in Fasting and OGTT 2h insulin and C-peptide levels
BMI, waist circumference, waist-to-hip ratio after 12weeks | Baseline , Day84
  Change from baseline in BMI, waist circumference, waist-to-hip ratio
Total body fat and visceral adipose tissue after 12weeks | Baseline , Day84
  Change from baseline in Total body fat and visceral adipose tissue
Blood lipid profile after 12weeks | Baseline , Day84
  Change from baseline in Blood lipid profile(include Triglycerides, total cholesterol, LDL-c, HDL-c)
TEAE and SAE | Up to 12 weeks
  Clinical significant Vital signs, physical and laboratory results

CONTACTS AND LOCATIONS:
Overall Officials: Yu Chen, Doctor, Principal Investigator — The Seventh Affiliated Hospital of Southern Medical University
Locations (1):
- The Seventh Affiliated Hospital of Southern Medical University, Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
In order to protect the privacy and security of the subject, the subject data will not be provided to other researchers